CLINICAL TRIAL: NCT01998022
Title: Hypertension of Our Patients: Knowledge, Control, Comorbidity
Acronym: H3C
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A00207-38; 651 (Other: CHM)
Record Dates: First submitted 2013-10-24; First posted 2013-11-28 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension
Keywords: hypertension; knowledge; blood pressure control
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Numerous studies highlight the insufficiency of blood pressure control in treated hypertensive population [1].

As shown in the MONICA study, increased cardiovascular mortality is found in Alsace compared to other french regions. The incidence and prevalence of diabetes and obesity are likely explanatory factors leading to this excess mortality [2].

Furthermore, the incidence and prevalence of alsacian patients with end-stage renal failure (ESRD) is also higher than the national average. The high prevalence of diabetes, hypertension and obesity in this population is also probably responsible for the high prevalence of ESRD [3].

Opportunities to prevent the progression of kidney disease involve an optimal control of treatable evolutionary factors.

Beyond control of diabetes and obesity, optimization of blood pressure control are an important factor to consider, as national and international guidelines recommend lower blood pressure targets in this population [4]. Knowledge of the disease and treatment goals are a key component of hypertensive patient management. Studies have shown that the knowledge of hypertensive disease and therapeutic targets were correlated with treatment compliance and with the rate of blood pressure control [5]. Patient education and participation of non-medical actors (nurses, pharmacists, …) are likely to improve the management and treatment compliance of these patients [6]. To our knowledge, no investigation has been performed in our region to determine the epidemiological characteristics, the knowledge level and blood pressure control in the population of hypertensive patients. The main objectives of this observational study are to evaluate, in a treated hypertensive population:

the knowledge level of the blood pressure treatment goals, the impact of patient knowledge on this blood pressure control, the potential impact of the patient's comorbidities on his blood pressure control.

Such a study should provide the basis for the feasibility of a large survey.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients moving spontaneously to their pharmacy to get their usual medications, including at least one drug in the class of anti-hypertensive

Exclusion Criteria:

* Refusal or inability of the patient to respond to the questionnaire.
* Antihypertensive therapy changed in the month preceding the survey.
* Antihypertensive therapy initiated within three months preceding the survey.
* Age <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treated hypertensive population
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
percentage of patients knowing the blood pressure target | Patients are included for the time of form completion, an expected average of 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- CHMulhouse, Mulhouse, France

REFERENCES:
- [Background] Mancia G, Sega R, Milesi C, Cesana G, Zanchetti A. Blood-pressure control in the hypertensive population. Lancet. 1997 Feb 15;349(9050):454-7. doi: 10.1016/s0140-6736(96)07099-7. PMID 9040574
- [Background] Berard E, Bongard V, Arveiler D, Amouyel P, Wagner A, Dallongeville J, Haas B, Cottel D, Ruidavets JB, Ferrieres J. Ten-year risk of all-cause mortality: assessment of a risk prediction algorithm in a French general population. Eur J Epidemiol. 2011 May;26(5):359-68. doi: 10.1007/s10654-010-9541-6. Epub 2010 Dec 28. PMID 21188478
- [Background] Registre REIN Rapport annuel 2010
- [Background] Mancia G, Laurent S, Agabiti-Rosei E, Ambrosioni E, Burnier M, Caulfield MJ, Cifkova R, Clement D, Coca A, Dominiczak A, Erdine S, Fagard R, Farsang C, Grassi G, Haller H, Heagerty A, Kjeldsen SE, Kiowski W, Mallion JM, Manolis A, Narkiewicz K, Nilsson P, Olsen MH, Rahn KH, Redon J, Rodicio J, Ruilope L, Schmieder RE, Struijker-Boudier HA, Van Zwieten PA, Viigimaa M, Zanchetti A. Reappraisal of European guidelines on hypertension management: a European Society of Hypertension Task Force document. Blood Press. 2009;18(6):308-47. doi: 10.3109/08037050903450468. No abstract available. PMID 20001654
- [Background] Atallah A, Papouin G, Mimran C, Braunstein C, Ganty J, Larifla L, Djaballah K, Inamo J. [Knowledge of hypertension among hypertensive patients in general practice, and its relation to achieving therapeutic goals: The Co-HACT study, French West Indies]. Ann Cardiol Angeiol (Paris). 2011 Feb;60(1):21-6. doi: 10.1016/j.ancard.2010.06.001. Epub 2010 Jul 16. French. PMID 20800218
- [Background] M Ashok Kumar. Improving medication adherence and clinical outcomes of hypertensive patients through patient counseling. Research Journal of Pharmaceutical, Biological and Chemical Sciences 2011; 2: 232-241